CLINICAL TRIAL: NCT02563522
Title: A Phase III, Double-blind, Randomized, Placebo-controlled, Multicenter Study to Assess the Safety and Efficacy of VM202 to Treat Chronic Nonhealing Foot Ulcers in Diabetic Patients With Concomitant Peripheral Arterial Disease (PAD)
Brief Title: Safety and Efficacy Study of Engensis (VM202) in the Treatment of Chronic Non-Healing Foot Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VMNHU-003
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Results first posted 2023-02-22 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-08

CONDITIONS: Foot Ulcer, Diabetic
Keywords: non healing ulcers; VM202; Diabetic ulcers; foot ulcers; Engensis
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Intervention Model Description: Active: Engensis (VM202) + standard of care - 200 subjects Control: Placebo (VM202 vehicle) + standard of care - 100 subjects
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Engensis (VM202) + standard of care
  Interventions: Genetic: Engensis (VM202)
- Control (Placebo Comparator): Placebo (VM202 Vehicle) + standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Genetic: Engensis (VM202) — gene therapy
  Arms: Active
Drug: Placebo — Standard of care plus placebo
  Other Names: VM202 vehicle
  Arms: Control

SUMMARY:
This study will assess the safety and efficacy of using gene therapy via intramuscular injections of the calf for patients with chronic non-healing foot ulcers.

DETAILED DESCRIPTION:
A phase III, randomized, double-blind, placebo-controlled, multicenter, 7-month study designed to assess the safety and efficacy of intramuscular (IM) injections in the calf of Engensis (VM202) in patients with chronic nonhealing foot ulcers. Three hundred patients will be randomized in a 2:1 ratio of VM202 or placebo injections:

* Active -Engensis (VM202) + standard of care - 200 patients
* Control - Placebo (VM202 Vehicle) + standard of care - 100 patients

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 80 years of age
2. Documented history of symptomatic PAD, with one or more of the following criteria satisfied:

   1. ABI >0.40 and ≤0.90 or >1.4 (i.e., mild to severe PAD without critical limb ischemia) in target limb
   2. TBI ≤0.7 in the target limb
   3. Toe pressure of <55 mmHg in the target limb
   4. A history of lower extremity PAD with previous related intervention in a leg
3. Documented history of Type I or II diabetes with current treatment control (HbA1c of ≤12.0% at Screening) and currently on oral medication, injectable medication, and/or insulin
4. No significant changes were anticipated in diabetes medication regimen
5. At Screening, the subject had one ulcer on the target foot that fulfilled all of the following criteria:

   1. Present for ≥2 weeks and ≤1 year
   2. Full-thickness and not involving bone, tendon, or capsule (probing to tendon or capsule)
   3. No sign of infection or osteomyelitis
   4. Ulcer must have been 0.5 cm2 to 15 cm2 as measured at the Screening visit prior to debridement If more than one ulcer was present on the foot, the largest ulcer that fulfilled the inclusion and exclusion criteria was considered the target (index) ulcer for the study. Subjects underwent protocol-defined standardized wound care during Screening (for two weeks or longer). Subjects were considered screen failures and did not receive study injections on Day 0 (Baseline) if the target ulcer did not meet all entry criteria (see above) as well as being confirmed as nonhealing.
6. Capable of understanding and complying with the protocol and signed the informed consent document prior to being subjected to any study related procedures
7. If female of childbearing potential, negative urine pregnancy test at Screening and used an acceptable method of birth control during the study

Exclusion Criteria:

1. Required revascularization in the target leg within 3 months of randomization
2. In the Investigator's assessment, required an amputation in the target leg within 3 months of randomization
3. Subjects with target foot ulcer with an etiology of vasculitis, pyoderma gangrenosum, necrobiosis lipoidica, hydrostatic pressure/venous insufficiency, any neoplasms (basalioma, Kaposi's sarcoma, squamous cell carcinoma, etc.), or due to a burn
4. The study ulcer increased or decreased by 50% or more at Baseline from Screening (as assessed by comparison of post-debridement photos taken at Screening and Day 0)
5. Evidence of active infection (e.g., cellulitis, osteomyelitis) or deep ulceration exposing bone or tendon in the foot planned for treatment
6. Any gangrene
7. Current fracture in the target foot
8. Target ulcer located on an active (hot) Charcot foot
9. Heart Failure with a New York Heart Association (NYHA) classification of III or IV
10. Body mass index (BMI) >45 kg/m2 at Screening
11. Stroke or myocardial infarction within the last 3 months
12. Unstable angina
13. Uncontrolled hypertension defined as sustained systolic blood pressure (SBP) >200 mmHg or diastolic blood pressure (DBP) >110 mmHg at Baseline/Screening evaluation
14. Ophthalmologic conditions pertinent to proliferative retinopathy or conditions that precluded standard ophthalmologic examination
15. Inflammatory disorder of the blood vessels (inflammatory angiopathy, such as Buerger's disease)
16. Subjects with advanced liver disease including decompensated cirrhosis, jaundice, ascites, or bleeding varices
17. Subjects currently receiving immunosuppressive medications chemotherapy, or radiation therapy
18. Positive human immunodeficiency virus (HIV) or human T-cell lymphotropic virus (HTLV) at Screening
19. Active hepatitis B or C infection as determined by hepatitis B surface antibody (HBsAb), hepatitis B core antibody (immunoglobulin G [IgG] and immunoglobulin M [IgM]; HBcAb), hepatitis B surface antigen (HBsAg), and hepatitis C antibodies (Anti-HCV) at Screening
20. Clinically significant specific laboratory values at Screening (e.g., hemoglobin <8.0 g/dL, white blood cell [WBC] <3,000/μL, platelet count <75,000/mm3, aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT] >3 times the upper limit of normal, or any other clinically significant lab abnormality which in the opinion of the Investigator was exclusionary)
21. Glomerular filtration rate (GFR) <30 mL/min/1.73 m2
22. Subjects with a recent history (<5 years) of or new Screening finding of malignant neoplasm except basal cell carcinoma or squamous cell carcinoma of the skin (if excised and no evidence of recurrence for at least 1 year); subjects with medical history and/or family history of colon cancer in any first degree relative were excluded unless they had undergone a colonoscopy in the last 12 months with negative findings
23. Subjects with any comorbid conditions likely to have interfered with assessment of safety or efficacy or with an estimated life expectancy of less than 1 year
24. Subjects who required >81 mg daily of acetylsalicylic acid. If >81 mg was taken at Screening, subjects could be enrolled if they were willing/able to switch to another medication for the duration of the study
25. Subjects who required regular (daily) COX-2 inhibitor drug(s) or steroids (except inhaled steroids or ocular steroids); subjects could be enrolled if they were willing/able to undergo medication washout prior to the first dosing and refrained from taking these drugs during the study
26. Major psychiatric disorder in the past 6 months
27. History of drug or alcohol abuse/dependence in the past 2 years
28. Used an investigational drug in the past 3 months; used an investigational biologic in the past 12 months; concurrent participation in an investigational protocol or using unapproved therapeutics
29. Was unable or unwilling to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emerson C. Perin, MD, Principal Investigator — Texas Heart Institute; David G Armstrong,, DPM, MD, PhD, Principal Investigator — Keck School of Medicine of University of Southern California
Locations (22):
- United States (22):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - NEA Baptist, Jonesboro, Arkansas
  - Sacramento Foot and Ankle, Carmichael, California
  - Bay Area Foot and Ankle, Castro Valley, California
  - VA Long Beach Healthcare System, Long Beach, California
  - USC Keck School of Medicine, Los Angeles, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Center for Clinical Research Inc., San Francisco, California
  - Olive View-UCLA Education & Research Institute, Sylmar, California
  - LCC Medical Research Institute, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - UMASS Memorial Med Center, Worcester, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Oregon Foot and Ankle Center, Eugene, Oregon
  - MedResearch, Inc, El Paso, Texas
  - Acclaim Bone & Joint Institute, Fort Worth, Texas
  - Texas Heart Institute, Houston, Texas
  - Futuro Clinical Trials, McAllen, Texas

REFERENCES:
- [Background] Perin E, Loveland L, Caporusso J, Dove C, Motley T, Sigal F, Vartivarian M, Oliva F, Armstrong DG; VMNHU-003 study group. Gene therapy for diabetic foot ulcers: Interim analysis of a randomised, placebo-controlled phase 3 study of VM202 (ENGENSIS), a plasmid DNA expressing two isoforms of human hepatocyte growth factor. Int Wound J. 2023 Nov;20(9):3531-3539. doi: 10.1111/iwj.14226. Epub 2023 May 25. PMID 37230802

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Control
Started | 27 | 17
Completed | 23 | 12
Not Completed | 4 | 5
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — withdrew consent,, noncompliance, and unable to attend future visits | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 27 | 17 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 8 | 28
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (11.05) | 61.2 (10.88) | 58.9 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 20 | 12 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 21 | 15 | 36
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 17 | 44

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With a Target Wound Closure by the 4-month Follow-up Visit
Description: Determine the proportion of subjects with a target Wound Closure from baseline to month 4 visit
Time Frame: Days 0 to Month 4
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 27 | 17
Participants | 13 | 5
Statistical Analysis 1: Comparison: Active vs Control; The statistical hypotheses were H0: Pt = Pc versus Ha: Pt ≠ Pc, where Pt and Pc are the proportions of subjects with a confirmed target would closure by the 4-month follow-up for Active (Engensis) and Control (Placebo) groups, respectively. The hypothesis testing was a two-sided alpha of 0.05; Test type: Other; p = 0.3455, Fisher Exact; No imputation was performed for subjects with missing response data; Mean Difference (Final Values) = 18.7, 95% CI 2-sided [-12.37 to 45.81]

ADVERSE EVENTS:
Time Frame: Day 0 to 7 months
Description: Treatment-emergent serious adverse events (TESAEs)
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/17
Serious Adverse Events (participants affected / at risk) | 11/27 | 5/17
Other Adverse Events (participants affected / at risk) | 16/27 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=27) | Control (N=17)
Infected skin ulcer (Infections and infestations) | 2 | 2
Osteomyelitis (Infections and infestations) | 4 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Hypoglycaemic encrephalopathy (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=27) | Control (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Blepharitis (Ear and labyrinth disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Macular oedema (Eye disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 6
Fungal infection (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 3 | 4
Influenza (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 2
Paronychia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 3 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 2
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 1
Glomerular filtration rate increased (Investigations) | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Hyperkalaemia (Investigations) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Exocytosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Mental status change (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 | 6
Haematoma (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02563522/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02563522/SAP_001.pdf